CLINICAL TRIAL: NCT06635993
Title: Accuracy of 68Ga-Pentixafor PET/CT for Subtypting Diagnosis in Patients With Primary Aldosteronism Concurrent With Autonomous Cortisol Secretion
Acronym: ABOARD
Status: Recruiting | Type: Observational
Sponsor: Qifu Li (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The Third Xiangya Hospital of Central South University (Other); The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Sponsor-Investigator, Qifu Li, Primary investigator, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Other Study IDs: ABOARD study
Record Dates: First submitted 2024-10-09; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Primary Aldosteronism Concurrent With Autonomous Cortisol Secretion
Keywords: primary aldosteronism; autonomous cortisol secretion; Adrenal venous sampling; 68Ga-Pentixafor PET/CT
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 68Ga-Pentixafor PET/CT — The patients had a normal diet with no special preparation before 68Ga-Pentixafor PET/CT imaging. The dosage of intravenously injected 68Ga-Pentixafor was calculated based on the patient's weight (1.85 MBq [0.05mCi]/kg). Local PET/CT scanning of the upper abdomen was performed on a hybrid PET/CT scanner at 10 minutes after the injection of the intravenous tracer, respectively.

SUMMARY:
To evaluate the accuracy of 68Ga-Pentixafor PET-CT in the classification diagnosis of primary aldosteronism concurrent with autonomous cortisol secretion patient, using AVS and/or postoperative remission as the reference standard for classification diagnosis.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, diagnostic trial involving patients with primary aldosteronism (PA) concurrent with autonomous cortisol secretion (ACS) patients with adrenal nodule (≥1cm) who completed both AVS and 68Ga-Pentixafor PET/CT. We will enroll 97 PA concurrent with ACS patients with adrenal nodule (≥1cm) .The treatment plan was determined according to the AVS results. AVS and/or postoperative remission were used as the reference standard for classification diagnosis to evaluate the accuracy of 68Ga-Pentixafor PET-CT in the classification diagnosis of PA concurrent with ACS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Getting the written informed consent
2. The clear diagnosis of primary aldosteronism；
3. Combined with autonomous cortisol secretion, cortisol after 1mg dexamethasone suppression test (DST) ≥50 nmol/l；
4. Patients who are willing to undergo surgery；
5. Adrenal CT or MRI scan of the adrenal glands with nodule (≥1cm).

Exclusion Criteria:

1. PA patients who meet the by-passing AVS criteria [i.e., younger than 35 years old, spontaneous hypokalemia, adrenal CT indicated unilateral low-density adenoma (≥1cm), plasma aldosterone >300pg/ml]；
2. Suspicion of familial hyperaldosteronism or Liddle syndrome. [i.e., age <20 years, hypertension and hypokalemia, or with family history]；
3. Suspicion of pheochromocytoma or adrenal carcinoma；
4. Patients with actively malignant tumor；
5. Patients who have adrenalectomy history；
6. Long-term use of glucocorticoids；
7. Patients who are allergic to contrast media and cannot tolerate AVS；
8. Pregnant or lactating women; with alcohol or drug abuse and mental disorders；
9. Congestive heart failure with New York Heart Association (NYHA) Functional Classification III or IV; History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 3 months; Severe anemia (Hb<60g/L); Serious liver dysfunction or chronic kidney disease aspartate aminotransferase (AST) or alanine transaminase (ALT) ≥3 times the upper limit of normal, or estimated glomerular filtration rate (eGFR) <30 ml/min/1.73 m2); Systemic Inflammatory Response Syndrome (SIRS); Uncontrolled diabetes (FBG≥13.3 mmol/L); Obesity (BMI≥35 kg/m²); Untreated aneurysm; Other comorbidity potentially interfering with treatment；
10. Consider patients with bilateral cortisol hypersecretion such as PBMAH or PPNAD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PA concurrent with ACS patients were from The First Affiliated Hospital of Chongqing Medical University, The Affiliated Hospital of Southwest Medical University, The Third Xiangya Hospital of Central South University, The First Affiliated Hospital of Zhengzhou University and Nanjing Drum Tower Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-08-12 (Estimated); Study Completion 2027-08-12 (Estimated)

PRIMARY OUTCOMES:
the accuracy of 68Ga-Pentixafor PET-CT in the classification diagnosis of PA concurrent with ACS patient | 6 months
  To evaluate the accuracy of 68Ga-Pentixafor PET-CT in the classification diagnosis of primary aldosteronism concurrent with autonomous cortisol secretion patient, using AVS and/or postoperative remission as the reference standard for classification diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Qi fu Li, PhD, Study Chair — the Chongqing Primary Aldosteronism Study (CONPASS) Group
Locations (1):
- The First Affilated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Libianto R, Russell GM, Stowasser M, Gwini SM, Nuttall P, Shen J, Young MJ, Fuller PJ, Yang J. Detecting primary aldosteronism in Australian primary care: a prospective study. Med J Aust. 2022 May 2;216(8):408-412. doi: 10.5694/mja2.51438. Epub 2022 Feb 25. PMID 35218017
- [Result] Xu Z, Yang J, Hu J, Song Y, He W, Luo T, Cheng Q, Ma L, Luo R, Fuller PJ, Cai J, Li Q, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Primary Aldosteronism in Patients in China With Recently Detected Hypertension. J Am Coll Cardiol. 2020 Apr 28;75(16):1913-1922. doi: 10.1016/j.jacc.2020.02.052. PMID 32327102
- [Result] Inoue K, Kitamoto T, Tsurutani Y, Saito J, Omura M, Nishikawa T. Cortisol Co-Secretion and Clinical Usefulness of ACTH Stimulation Test in Primary Aldosteronism: A Systematic Review and Biases in Epidemiological Studies. Front Endocrinol (Lausanne). 2021 Mar 16;12:645488. doi: 10.3389/fendo.2021.645488. eCollection 2021. PMID 33796078
- [Result] Buffolo F, Pieroni J, Ponzetto F, Forestiero V, Rossato D, Fonio P, Nonnato A, Settanni F, Mulatero P, Mengozzi G, Monticone S. Prevalence of Cortisol Cosecretion in Patients With Primary Aldosteronism: Role of Metanephrine in Adrenal Vein Sampling. J Clin Endocrinol Metab. 2023 Aug 18;108(9):e720-e725. doi: 10.1210/clinem/dgad179. PMID 36974473
- [Result] Spath M, Korovkin S, Antke C, Anlauf M, Willenberg HS. Aldosterone- and cortisol-co-secreting adrenal tumors: the lost subtype of primary aldosteronism. Eur J Endocrinol. 2011 Apr;164(4):447-55. doi: 10.1530/EJE-10-1070. Epub 2011 Jan 26. PMID 21270113
- [Result] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Result] Naruse M, Katabami T, Shibata H, Sone M, Takahashi K, Tanabe A, Izawa S, Ichijo T, Otsuki M, Omura M, Ogawa Y, Oki Y, Kurihara I, Kobayashi H, Sakamoto R, Satoh F, Takeda Y, Tanaka T, Tamura K, Tsuiki M, Hashimoto S, Hasegawa T, Yoshimoto T, Yoneda T, Yamamoto K, Rakugi H, Wada N, Saiki A, Ohno Y, Haze T. Japan Endocrine Society clinical practice guideline for the diagnosis and management of primary aldosteronism 2021. Endocr J. 2022 Apr 28;69(4):327-359. doi: 10.1507/endocrj.EJ21-0508. Epub 2022 Apr 12. PMID 35418526
- [Result] Rossi GP, Bisogni V, Bacca AV, Belfiore A, Cesari M, Concistre A, Del Pinto R, Fabris B, Fallo F, Fava C, Ferri C, Giacchetti G, Grassi G, Letizia C, Maccario M, Mallamaci F, Maiolino G, Manfellotto D, Minuz P, Monticone S, Morganti A, Muiesan ML, Mulatero P, Negro A, Parati G, Pengo MF, Petramala L, Pizzolo F, Rizzoni D, Rossitto G, Veglio F, Seccia TM. The 2020 Italian Society of Arterial Hypertension (SIIA) practical guidelines for the management of primary aldosteronism. Int J Cardiol Hypertens. 2020 Apr 15;5:100029. doi: 10.1016/j.ijchy.2020.100029. eCollection 2020 Jun. PMID 33447758
- [Result] Kline GA, Dias VC, So B, Harvey A, Pasieka JL. Despite limited specificity, computed tomography predicts lateralization and clinical outcome in primary aldosteronism. World J Surg. 2014 Nov;38(11):2855-62. doi: 10.1007/s00268-014-2694-9. PMID 25002246
- [Result] Sam D, Kline GA, So B, Leung AA. Discordance Between Imaging and Adrenal Vein Sampling in Primary Aldosteronism Irrespective of Interpretation Criteria. J Clin Endocrinol Metab. 2019 Jun 1;104(6):1900-1906. doi: 10.1210/jc.2018-02089. PMID 30590677
- [Result] Young WF, Stanson AW, Thompson GB, Grant CS, Farley DR, van Heerden JA. Role for adrenal venous sampling in primary aldosteronism. Surgery. 2004 Dec;136(6):1227-35. doi: 10.1016/j.surg.2004.06.051. PMID 15657580
- [Result] Kuil J, Buckle T, van Leeuwen FW. Imaging agents for the chemokine receptor 4 (CXCR4). Chem Soc Rev. 2012 Aug 7;41(15):5239-61. doi: 10.1039/c2cs35085h. Epub 2012 Jun 28. PMID 22743644
- [Result] Ding J, Tong A, Hacker M, Feng M, Huo L, Li X. Usefulness of 68 Ga-Pentixafor PET/CT on Diagnosis and Management of Cushing Syndrome. Clin Nucl Med. 2022 Aug 1;47(8):669-676. doi: 10.1097/RLU.0000000000004244. Epub 2022 Apr 22. PMID 35452014
- [Result] Heinze B, Fuss CT, Mulatero P, Beuschlein F, Reincke M, Mustafa M, Schirbel A, Deutschbein T, Williams TA, Rhayem Y, Quinkler M, Rayes N, Monticone S, Wild V, Gomez-Sanchez CE, Reis AC, Petersenn S, Wester HJ, Kropf S, Fassnacht M, Lang K, Herrmann K, Buck AK, Bluemel C, Hahner S. Targeting CXCR4 (CXC Chemokine Receptor Type 4) for Molecular Imaging of Aldosterone-Producing Adenoma. Hypertension. 2018 Feb;71(2):317-325. doi: 10.1161/HYPERTENSIONAHA.117.09975. Epub 2017 Dec 26. PMID 29279316
- [Result] Hu J, Xu T, Shen H, Song Y, Yang J, Zhang A, Ding H, Xing N, Li Z, Qiu L, Ma L, Yang Y, Feng Z, Du Z, He W, Sun Y, Cai J, Li Q, Chen Y, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Accuracy of Gallium-68 Pentixafor Positron Emission Tomography-Computed Tomography for Subtyping Diagnosis of Primary Aldosteronism. JAMA Netw Open. 2023 Feb 1;6(2):e2255609. doi: 10.1001/jamanetworkopen.2022.55609. PMID 36795418